CLINICAL TRIAL: NCT06234202
Title: The Effect of a Bioactive Fabric Sleeve on Recovery in Division I Collegiate Baseball Players
Brief Title: The Effect of a Bioactive Fabric Sleeve
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Challenger Health, LLC (Unknown)
Responsible Party: Principal Investigator, Michael T. Freehill, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 72979
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Recovery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bioactive Sleeve then Control Sleeve (Experimental): Each pitcher will be instructed to sleep with the assigned sleeve on the throwing arm after each game that he pitches
  Interventions: Device: Bioactive Sleeve; Device: Control Sleeve
- Control Sleeve then Bioactive Sleeve (Experimental): Each pitcher will be instructed to sleep with the assigned sleeve on the throwing arm after each game that he pitches
  Interventions: Device: Bioactive Sleeve; Device: Control Sleeve

INTERVENTIONS:
Device: Bioactive Sleeve — Pitchers will wear a bioactive sleeve immediately post-game through overnight.
Device: Control Sleeve — Pitchers will wear a non-bioactive sleeve immediately post-game through overnight.

SUMMARY:
In-season pitch volume have been shown to relate to arm soreness in collegiate baseball players. Arm soreness is a common ailment following a pitching appearance due to the adaptation to soft tissue in response to a repetitive load to the throwing arm. Specifically, ongoing and accumulated fatigue and soreness to the flexor pronator mass region of the arm may be a predecessor for UCL injury. Different recovery modalities such as a bioactive fabric sleeve may give pitchers a recovery advantage throughout a baseball season. The primary purpose of this study is to determine if there is a difference in subjective soreness of the flexor pronator mass the day following a game pitching appearance using a sleeve with bioactive fabric which potentially improves cellular function versus a control sleeve.

ELIGIBILITY:
Inclusion Criteria:

* Stanford Baseball Player

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Subjective Soreness Score | Baseline through 6 months
  Subjective soreness questionnaires to rank soreness, tightness, and discomfort of the medial forearm on a 1 to 10 scale will be collected throughout the baseball seasons.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Freehill, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No